CLINICAL TRIAL: NCT02642536
Title: Improving Obesity Self-care Among Mentally Ill Veterans
Acronym: MH MOVE!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7886-W
Record Dates: First submitted 2015-12-10; First posted 2015-12-30 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Anxiety; Depression; PTSD; Obesity
Keywords: Veteran
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking was Double Blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- MH MOVE (Active Comparator): provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms to be used during 10 phone based clinician led CBT sessions
  Interventions: Behavioral: MH MOVE
- Enhanced Usual Care (Active Comparator): provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms but not phone calls are provided.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: MH MOVE — provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms to be used during 10 phone based clinician led CBT sessions
  Arms: MH MOVE
Behavioral: Enhanced Usual Care — provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms but not phone calls are provided.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to find out which of two programs, MH MOVE! or the enhanced usual care MOVE! program is most effective in improving participation in and completion of MOVE! among Veterans with depression, anxiety, and PTSD. One of the treatments, MH MOVE! provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms to be used during 10 phone based clinician led CBT sessions. The enhanced usual care MOVE! provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms but not phone calls are provided.

DETAILED DESCRIPTION:
First-time, newly enrolled participants in the MOVE! program will be targeted for treatment. Recruitment will take place utilizing flyers and MEDVAMC clinician referral. The research coordinator, PI or other study staff will attend the MOVE! assessment group and individual MOVE! sessions. During this initial contact, a recruitment letter will be read to all potential subjects. The letter will provide an overview of the study and allow potential participants the opportunity to express interest in the study. Those who are interested will be invited to sign their name to a sheet indicating their interest in the study and their willingness to undergo the initial screening for eligibility. In order to determine eligibility, patient records will be accessed for inclusion and exclusion information. Veterans who meet the inclusion criteria will be contacted to schedule a time to sign the necessary consent forms and receive the pre-treatment screening assessment forms. The pre-treatment assessment will be conducted face to face and last approximately 1 hour. During this time, the research coordinator or other study staff will review the VA consent, VA 10-3203 consent to voice recording, and VA HIPPA forms and answer any additional questions. After all questions regarding consent and study enrollment are answered, the RC or other study staff will instruct the participant to sign the consent forms. The participants will receive hard copies of the VA consent, VA 10-3203 consent to voice recording, and VA HIPPA forms that contain all required signatures. The Veteran will then be provided the intake assessment forms. These forms will gather demographic data such as age, gender, ethnicity, race, education, marital status, employment, VA disability, and military history. Veterans will be asked about medications, other therapies, and hospitalizations. Additional screening assessments will measure mental health diagnosis and symptom severity. Veterans who continue to meet the inclusion criteria will then be included into the study. Veterans who do not meet the inclusion criteria but demonstrate a need or ask for additional services from the MEDVAMC will be referred for mental health care. In the randomized controlled trial, once Veterans have been consented, they will be randomized to the MH MOVE or enhanced usual-care MOVE! treatment group. Those who are randomized to the MH MOVE! group will be administered the 6 core, 2 optional, and 2 booster depression, anxiety and PTSD focused MH MOVE! treatment module sessions via phone.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be Veterans over 18 years of age who are overweight or obese as indicated by a BMI greater than 30.
* Participants who are enrolled have never participated in the MOVE! program and are joining the MOVE! program for the first time.
* Severity of potential co-existing anxiety and depression will be assessed by a diagnosis of PTSD, anxiety and depression noted in the medical history and will be confirmed using the PTSD Checklist (PCL-C), Patient Health Questionnaire (PHQ-8), Generalized Anxiety 7-item Scale (GAD-7).
* Participants who endorse mild-to-moderate depression characterized by a scores in the range of 5-19 on the PHQ-8, scores ranging from 5-14 on the GAD-7 scale and scores 6-50 on the PCL.

Exclusion Criteria:

* Participants will be excluded if they have a medical diagnosis of schizophrenia or bi-polar
* Have symptom checklist score in the severe range of anxiety, depression or PTSD
* Demonstrate suicidal/homicidal plan and intent
* And/or demonstrate moderate or severe cognitive impairment as demonstrated by the cognitive status screener
* Do not have regular access to a telephone
* Are no longer obese as established by calculation of current BMI
* Or are no longer endorsing any symptoms of anxiety or depression as established by a score of less than 5 (due to lack of depressive symptoms) and those greater than 19 (due to severity of depressive symptoms) on the PHQ-8 and less than 5 (indicating no presence of anxiety) and greater than 15 (indicating severe anxiety) on the GAD-7 less than 6 (indicating no presence of PTSD symptoms) and greater than 50 (severe PTSD) on the PCL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Evans, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MH MOVE | Enhanced Usual Care
Started | 21 | 23
Completed | 19 | 18
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- MH MOVE: provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms to be used during 8 phone based clinician led CBT sessions
  MH MOVE: provides the standard MOVE! weight management program plus a workbook containing education for management of depression, anxiety and PTSD symptoms to be used during 8 phone based clinician led CBT sessions
- Total: Total of all reporting groups
Arm/Group | MH MOVE | Enhanced Usual Care | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.65 (8.9) | 58.3 (9.5) | 58.65 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 19 | 20 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 12 | 20
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MOVE! Attendance
Description: Number of MOVE! sessions attended minimum-maximum total score range (2-12) Higher value represents more sessions attended The score was obtained from a single item
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: number of sessions
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
number of sessions | 5.9 (1.8) | 5.8 (1.8)

2. Primary Outcome: Number of Days Engaged in Vigorous Activity
Description: changes in vigor and time spent on physical activity practice will be measured by the MOVE! 11 assessment at post treatment (16 weeks) minimum-maximum total score range (0-48) Higher value represents more days spent performing vigorous activity
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: days spent performing vigorous activity
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
days spent performing vigorous activity | 21.5 (11.5) | 26.9 (18)

3. Primary Outcome: Number of Days Engaged in Vigorous Activity
Description: Initial assessment of vigor and time spent on physical activity minimum-maximum total score range (0-32) Higher value represents more days spent performing vigorous physical activity The score was obtained from a single item
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: days spent performing vigorous activity
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
days spent performing vigorous activity | 27.7 (22.1) | 28.1 (15.3)

4. Primary Outcome: Self Efficacy for Practicing Good Dietary Habits
Description: Self-efficacy for practicing healthy dietary habits during difficult times will be assessed at baseline and post treatment (16 weeks) minimum-maximum total score range (20-100) Higher value represents greater sense of self-efficacy for healthy eating during difficult times The score was obtained from 3 subscales
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 32.3 (19.2) | 29.8 (6.0)

5. Primary Outcome: Self Efficacy for Practicing Good Dietary Habits
Description: as for outcome 4
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 29.9 (10.4) | 23.2 (7.4)

6. Secondary Outcome: Assessing Depression Symptom Severity
Description: Changes in depression symptom severity will be measured at baseline and post treatment (16 weeks) minimum-maximum total score range (0-24) Higher value represents greater depressive symptom severity An overall score was obtained from the 8-item measure.
Time Frame: 16 weeks
Population: frequency analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 6.3 (7.1) | 13.4 (6.2)

7. Secondary Outcome: Assessing Anxiety Symptom Severity
Description: Anxiety symptom severity will be measured by the GAD-7 at baseline and post treatment (16 weeks) minimum-maximum total score range (0-21) Higher value represents greater anxiety symptom severity An overall score was obtained from the 7-item measure.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 5.5 (6.5) | 10.5 (6.7)

8. Secondary Outcome: Assessing PTSD Symptom Severity
Description: PTSD symptom severity will be measured by the PCL-M at baseline and post treatment (16 weeks) minimum-maximum total score range (17-85) Higher value represents greater PTSD symptom severity An overall score was obtained from 4 subscales.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 32.1 (20.8) | 53 (18)

9. Secondary Outcome: Assessing Depression Symptom Severity
Description: as for outcome 6
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 19 (21.7) | 15 (19.3)

10. Secondary Outcome: Assessing Anxiety Symptom Severity
Description: as for outcome 7
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 8 (13.8) | 16 (19.7)

11. Secondary Outcome: Assessing PTSD Symptom Severity
Description: as for outcome 8
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MH MOVE | Enhanced Usual Care
Number analyzed (Participants) | 19 | 18
units on a scale | 39 (26.5) | 25 (73.5)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected during the entire 2 year study time frame.
Arm/Group | MH MOVE | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes